CLINICAL TRIAL: NCT01616238
Title: A Phase 2 Study for Older Adults With Acute Lymphoblastic Leukaemia
Brief Title: A Study for Older Adults With Acute Lymphoblastic Leukaemia
Acronym: UKALL60+
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/11/0532
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Acute Lymphoblastic Leukaemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Philadelphia Positive Patients (Experimental): All patients with Philadelphia positive ALL will be treated in this group and will receive a standard imatinib-containing chemotherapy regimen
  Interventions: Drug: Chemotherapy
- Philadelphia -ve Patients- Intensive (Experimental): Patients with Philadelphia negative ALL who are fit for intensive treatment will be allocated into this group.
  Interventions: Drug: Chemotherapy
- Philadelphia -ve Patients- Intensive + (Experimental): Patients with Philadelphia negative disease and who are fit for intensive treatment will be entered into this group
  Interventions: Drug: Chemotherapy
- Philadelphia -ve Patients- Non Intensive (Experimental): Patients with Philadelphia negative disease who are not fit for intensive chemotherapy will be entered into this group
  Interventions: Drug: Chemotherapy
- Registration only (No Intervention): Patients with either Philadelphia positive or negative ALL who do not wish to enter the study will be allocated to this group for data collection purposes only.

INTERVENTIONS:
Drug: Chemotherapy — Treatment for all pathways consists of Induction, Intensification (where applicable), Consolidation and Maintenance therapy during which combination chemotherapy is given for up to 2.5 years.
  Arms: Philadelphia -ve Patients- Intensive; Philadelphia -ve Patients- Intensive +; Philadelphia -ve Patients- Non Intensive; Philadelphia Positive Patients

SUMMARY:
The NCRI Adult ALL sub-group propose to collaborate with the Dutch/Belgian group HOVON to carry out a prospective, non randomised multi-arm study (including a choice of regimen intensity) to investigate the safety, tolerability and feasibility of a standardised therapy protocol for patients ≥ 60 years old with de novo ALL. The overall aim is define a basic standard of care upon which trials of novel therapies will be based in future. The design of the study will enable collection of a comprehensive dataset regarding the clinical outcome, Complete Response Rate (CR) and Minimal Residual Disease (MRD) response rates in a previously completely uncharacterised population, thus providing the essential platform for designing future randomised advanced phase studies in which new therapeutic approaches and novel therapies can be prospectively investigated.

DETAILED DESCRIPTION:
The study will

1. establish baseline expectations for Event Free Survival (EFS), Overall Survival (OS), MRD responses and quality of life measures for older patients of all ages and pre-morbid states;
2. disclose how best to use knowledge of pre-morbid characteristics to apply the appropriate intensity of therapy in order to balance the best disease related outcomes against quality of life;
3. establish national standards of care for this patient group;
4. provide the essential platform for careful design of future randomised advanced phase studies of new therapeutic approaches and agents.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 with Acute Lymphoblastic Leukaemia (ALL) OR ≥ 55 with Acute Lymphoblastic Leukaemia (ALL) unsuitable for the UKALL14 or HOVON 100 trial
* Newly diagnosed, previously untreated ALL (a steroid pre-phase of 5-7 days may be given before trial registration))
* Willing and able to give consent

Exclusion Criteria:

* Known HIV infection
* Blast transformation of CML
* Mature B-cell leukaemia i.e. Burkitts disease t(8,14)(q24 ;q32) and variant c-myc translocations e.g. t(2;8)(p12 ;q24), t(8;22)(q24;q11)
* Women who are pregnant or lactating

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-12; Primary Completion 2018-12-21 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Complete remission rate after 2 phases of induction | Approximately 2 months after start of treatment
  All patients will be assessed for their remission status at the end of Phase 2 induction. The CR rate at this timepoint will then be calculated.

SECONDARY OUTCOMES:
Complete remission rate after 1 phase of induction | Approximately 1 month after start of treatment
  All patients will be assessed for their remission status at the end of Phase 1 induction. The CR rate at this timepoint will then be calculated.
Overall Survival at 1 year | 1 year after registration
  Overall survival for all patients will be measured 1 year after registration
Prognostic significance of molecularly determined minimal residual disease (MRD) at various time-points during therapy with respect to relapse occurrence. | At diagnosis, 4 weeks, 8 weeks, 12 weeks after starting treatment
  MRD levels will be measured at distinct timepoints during the trial.
Tolerability of treatment as determined by occurrence of key adverse effects | Approximately 4 weeks, 8 weeks, 12 weeks, 24 weeks after starting treatment
  Patients in arms A-D will be assessed for adverse events at distinct timepoints during the trial
Duration of in-patient hospitalisation | Approximately 4 weeks, 8 weeks, 12 weeks, 24 weeks, 28 after starting treatment and every 3 months during maintenance
  All patients will be assessed for the number of days they have spent as in-patients at distinct timepoints during the trial.
Relationship between performance status/co-morbidity and treatment option chosen | At registration
Quality of life aspects assessed at diagnosis/baseline at various time points | Registration, Approximately 4 weeks, 8 weeks, 12 weeks, 24 weeks, 28 after starting treatment, before starting maintenance and at the end of maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Prof Adele Fielding, Principal Investigator — University College London Hospital
Locations (34):
- Erasmus MC, Rotterdam, Netherlands
- United Kingdom (33):
  - NHS Lanarkshire - Monklands, Airdrie
  - Blackpool Victoria Hopsital, Blackpool
  - Royal Bournemouth Hospital, Bournemouth
  - Bradford Royal Infirmary, Bradford
  - Bristol Haematology and Oncology Centre, Bristol
  - University Hospital of Wales, Cardiff
  - Castle Hill Hospital, Cottingham
  - Russells Hall Hospital, Dudley
  - Ninewells Hospital, Dundee
  - NHS Lothian - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - New Victoria Hospital and Southern General Hospital, Glasgow
  - Northwick Park Hospital, Harrow
  - St James' Hospital, Leeds, Leeds
  - Leicester Royal Infirmary, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - King's College Hospital NHS Foundation Trust, London
  - St Bartholomew's Hospital, London
  - St George's Hospital, London
  - The Christie Hospital, Manchester
  - Arrowe Park Hospital, Metropolitan Borough of Wirral
  - James Cook University Hospital, Middlesbrough
  - Churchill Hospital, Oxford, Oxford
  - Derriford Hospital, Plymouth
  - Poole General Hospital, Poole
  - St Helen's & Knowlsey Teaching Hospitals, Prescot
  - Salisbury District Hospital, Salisbury
  - Royal Hallamshire Hospital, Sheffield
  - Royal MarsdenHospital, Sutton
  - Great Western Hospital, Swindon
  - Musgrove Park, Taunton
  - Torbay Hospital, Torquay
  - Sandwell General Hospital, West Bromwich